CLINICAL TRIAL: NCT01918215
Title: Cardiac Magnetic Resonance GUIDEd Management of Mild-moderate Left Ventricular Systolic Dysfunction
Acronym: CMR_GUIDE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Flinders University (Other)
Collaborators: South Australian Health and Medical Research Institute (Other)
Responsible Party: Principal Investigator, Joseph Selvanayagam, Professor Joseph Selvanayagam, Flinders University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CMRG-HF-1
Record Dates: First submitted 2013-04-19; First posted 2013-08-07 (Estimated); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Heart Failure; Left Ventricular Systolic Dysfunction
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction, Left

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Device Implantation (Other): A prospective, blocked, randomised, placebo-controlled trial of primary prophylaxis ICD therapy or implantable loop recorder (ILR) insertion in patients with LVEF 36-50% and Late Gadolinium Enhancement(LGE)on CMR
  Interventions: Device: ICD; Device: ILR
- Observational Registry (No Intervention): A prospective observational registry of patients with LVEF 36-50% and no LGE on CMR

INTERVENTIONS:
Device: ICD
  Arms: Device Implantation
Device: ILR
  Arms: Device Implantation

SUMMARY:
Contemporary heart failure (HF) guidelines recommend insertion of a primary prevention implantable defibrillator (ICD) in patients with left ventricular ejection fraction less than 35% (LVEF < 35%) on maximally tolerated medical therapy. Nevertheless, there are a substantial number of HF patients who have LVEF>35% and hence do not qualify for ICD, who succumb to sudden cardiac death (SCD). At present our tools to reliably risk stratify these patients with mild-moderate systolic dysfunction (LVEF 36-50%) are poor. It is likely that these patients have ventricular scar and/or replacement fibrosis as a substrate for their malignant arrhythmia. Cardiovascular magnetic resonance imaging (CMR) can reliably identify and quantify both ventricular scar (seen in Ischaemic cardiomyopathy, ICM) and replacement myocardial fibrosis (seen in Non-Ischemic Cardiomyopathy, NICM).

Methods/Design: A multi-centre randomised controlled trial in which 428 patients with mild-moderate left-ventricular systolic dysfunction (either ICM or NICM) and ventricular scar/fibrosis on cardiovascular magnetic resonance are randomized to either ICD or implantable loop recorder (ILR) insertion and are followed up until the last patient recruited has been in the study for 3 years.

Potentially eligible patients will have a screening CMR and will be enrolled into the device arm of study based on the presence of any ventricular scar/fibrosis (CMR +). Patients who do not have ventricular scar/fibrosis will be followed up in an observational registry, and will not be randomised.

In both the device and registry arms, we aim to enrol 700 patients in Australia and 355 in Europe.

The primary hypothesis is that among patients with mild-moderate left ventricular systolic dysfunction, a routine CMR guided management strategy of ICD insertion is superior to a conservative strategy of standard care.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or greater than 18 years
* Patients with coronary artery disease (CAD) or dilated cardiomyopathy (DCM) of the idiopathic, chronic post myocarditis or familial type.
* Left ventricular systolic impairment as defined by left ventricular ejection fraction 36-50% by any current standard technique (echocardiogram, multiple gated acquisition scan (MUGA), angiography or CMR taken in the last six months. If a LGE CMR has been taken within 2 months this scan can be used for inclusion
* Able and willing to comply with all pre-, post- and follow-up testing, and requirements
* On maximum tolerated doses of ACE inhibitors (or Angiotensin and Receptor Blockers if intolerant of ACE) and Beta Blockers

Exclusion Criteria:

1. History of cardiac arrest or spontaneous or inducible sustained ventricular tachycardia or ventricular fibrillation unless within 48 hours of an acute MI
2. Cardiomyopathy related to sarcoidosis
3. Standard Cardiac Magnetic Resonance imaging contraindications (e.g. severe claustrophobia)
4. Currently implanted permanent pacemaker and/or pacemaker/ICD lead
5. Clinical indication for ICD or Pacemaker or cardiac resynchronisation therapy.
6. CMR LVEF ≤35% or>50%
7. Severe renal insufficiency (eGFR< 30mls/min/1.73m2)
8. Recent Myocardial Infarction (MI) (<40 days) or cardiac revascularization (<90 days)
9. New York Heart Association HF functional class IV at baseline
10. Conditions associated with life expectancy <1 year
11. Pregnancy or in females of child-bearing potential, the non-use of accepted forms of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Composite of Sudden Cardiac Death or haemodynamically significant ventricular arrhythmia | Through to study completion, an average of 4 years
  Defined as: ventricular arrhythmia producing syncope (loss of consciousness) or associated with hypotension (SBP<90mmHg) except directly associated with device implant procedure.

SECONDARY OUTCOMES:
Sudden Cardiac Death | Through to study completion, an average of 4 years
Haemodynamically significant ventricular arrhythmia | Through to study completion, an average of 4 years
All-cause mortality | Through to study completion, an average of 4 years
Change in New York Heart Association Functional class | 3, 6,12, 24, 36, 48 months
Heart failure related hospitalizations | Through to study completion, an average of 4 years
Health economic evaluation of cost | At study completion, average of 4 years
  Australia only
Quality of life assessed by Minnesota Living with Heart Failure Questionnaire | 3, 6,12, 24, 36, 48 months
Quality of life assessed by EuroQol-5D-5L questionnaire | 3, 6,12, 24, 36, 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Joseph B Selvanayagam, MBBS, Principal Investigator — Flinders Medical Centre
Locations (18):
- Australia (10):
  - John Hunter Hospital, New Lambton, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - St Vincent's Hospital, Fitzroy, Victoria
  - The Alfred, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Germany (3):
  - Coburg Hospital, Coburg
  - Schwarzwald-Baar Klinikum, Villingen-Schwenningen
  - University Hospital Wurzburg, Würzburg
- United Kingdom (5):
  - Belfast Health and Social Care Trust, Belfast
  - The Bristol Heart Institute, Bristol
  - Golden Jubilee National Hospital, Clydebank
  - Glenfield General Hospital, Leicester
  - University Hospital of South Manchester NHS Foundation Trust, Manchester

REFERENCES:
- [Derived] Selvanayagam JB, Hartshorne T, Billot L, Grover S, Hillis GS, Jung W, Krum H, Prasad S, McGavigan AD. Cardiovascular magnetic resonance-GUIDEd management of mild to moderate left ventricular systolic dysfunction (CMR GUIDE): Study protocol for a randomized controlled trial. Ann Noninvasive Electrocardiol. 2017 Jul;22(4):e12420. doi: 10.1111/anec.12420. Epub 2017 Jan 24. PMID 28117536